CLINICAL TRIAL: NCT00516880
Title: Targeting Peroxisome Proliferator-activated Receptor-gamma in Peritoneal Dialysis Patients - Will it Reduce Inflammation, Atherosclerosis, Calcification and Improve Survival of Peritoneal Dialysis Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW05-236T/899; HARECCTR0500007
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Disease; Kidney Diseases; Cardiovascular Diseases
Keywords: chronic kidney disease; cardiovascular disease
MeSH Terms: conditions — Chronic Disease; Kidney Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
Peritoneal dialysis patients are at increased risk of cardiovascular morbidity and mortality and are related to the presence of accelerated atherosclerosis. Our recent data showed that inflammation predicts mortality and cardiovascular death, independent of other cardiovascular risk factors in peritoneal dialysis patients. As a considerable proportion of peritoneal dialysis patients showed evidence of inflammation, it raises an important question as to whether anti-inflammatory treatment has any cardiovascular and survival benefit in these patients. The peroxisome proliferator-activated receptor-gamma (PPAR-g) agonist is a class of drug with insulin sensitizing property. Recent experimental and clinical studies demonstrated that this class of drug has anti-inflammatory and anti-atherosclerotic properties other than insulin sensitizing effect in type 2 diabetics. We therefore hypothesize that modulation of the PPAR-g activity may be a novel therapeutic strategy for reducing inflammation and retarding the progression of atherosclerosis and possibly lowering mortality in our peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Both prevalent patients or patients newly started on continuous ambulatory peritoneal dialysis with age between 20 - 75 with or without diabetes mellitus will be considered eligible for study entry. For patients newly started on continuous ambulatory peritoneal dialysis, they will be suitable for recruitment into the study after one month on continuous ambulatory peritoneal dialysis.

Exclusion Criteria:

* Patients with underlying malignancy
* Patients with chronic liver disease or liver cirrhosis
* Patients with hepatitis B or C positive
* Patients with active infections
* Patients with other chronic active inflammatory disease such as systemic lupus erythematosus, rheumatoid arthritis
* Patients who refuse study participation
* Patients with underlying congenital heart disease or rheumatic heart disease
* Patients with poor general condition
* Patients with plans for living related kidney transplant within 2 years
* Female patients with pregnancy
* Patients with history of recurrent hypoglycemia
* Patients with Class III and IV congestive heart failure
* Patients already receiving glitazones treatment at the screening visit

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-03; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
carotid athersclerosis | 6 month, 1 year and 2 year
endothelial function | 6 month, 1 year and 2 year

SECONDARY OUTCOMES:
all-cause mortality and cardiovascular event | 1 year, 2 year
pulse wave velocity | 6 month, 1 year, 2 year
inflammation | 6 month, 1 year, 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Angela Wang, Dr, Principal Investigator — Department of Medicine/Nephrology, Queen Mary Hospital/ The University of Hong Kong
Locations (2):
- China (2):
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Department of Medicine, Tung Wah Hospital, Hong Kong